CLINICAL TRIAL: NCT04659720
Title: Clinical Evaluation of Stability of Dental Implant Placed Simultaneously With Closed Sinus Lifting Using Hydraulic Lift Technique Versus Summer's Osteotome Technique in Posterior Edentulous Maxilla (Randomized Clinical Trial)
Brief Title: Clinical Evaluation of Stability of Dental Implant Placed Simultaneously With Closed Sinus Lifting Using Hydraulic Lift Technique Versus Summer's Osteotome Technique in Posterior Edentulous Maxilla (RCT)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hassan Mohammad, Assoc.professor in maxillo facial surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 131020
Record Dates: First submitted 2020-11-19; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Evaluations, Diagnostic Self

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- summers' osteotome technique for closed sinus lift (Active Comparator): Implant stability will be evaluated after closed sinus lift using summer's osteotome technique in posterior edentulous maxilla
  Interventions: Device: Hydrolic lifter device
- Patient satisfaction evaluation after closed sinus lifting using summers' osteotome technique (Active Comparator): * Will be assessed numerically using a patient satisfaction chart .
  * Time of assessment: immediately after surgery
  Interventions: Behavioral: Patient satisfaction evalution using hydraulic lifter device

INTERVENTIONS:
Device: Hydrolic lifter device — evaluation of implant stability after closed sinus lifting by hydraulic lift technique using hydraulic lifter device
  Arms: summers' osteotome technique for closed sinus lift
Behavioral: Patient satisfaction evalution using hydraulic lifter device — patients satisfaction will be evaluated numerically after using hydraulic lift technique by hydraulic lifter device for closed sinus lifting in posterior edentulous maxilla
  Arms: Patient satisfaction evaluation after closed sinus lifting using summers' osteotome technique

SUMMARY:
Clinical evaluation of stability of dental implant placed simultaneously with closed sinus lifting using hydraulic lift technique versus summer's osteotome technique in posterior edentulous maxilla (RCT)

DETAILED DESCRIPTION:
Clinical evaluation of stability of dental implant placed simultaneously with closed sinus lifting using hydraulic lift technique versus summer's osteotome technique in posterior edentulous maxilla (Randomised clinical trial)

ELIGIBILITY:
Inclusion Criteria:

* Edentulous patients in the maxillary posterior region.
* Patients in need to fixed restorations in posterior region.
* Patients with healthy systemic conditions. (Apparently medically free)
* Patients with adequate inter-arch space for placement of the prosthetic part of the implant .
* Patients who had approximately 5-8 mm of available bone height between crest of bone and floor of sinus
* Both sexes.
* Patients with Good oral hygiene
* Patients more than 20 years old
* Cooperative and motivated patients

Exclusion Criteria:

* Patients with local pathological defects related to posterior maxilla.
* Heavy smokers.
* Abnormal habits that may alter results such as alcoholism or parafunctional habits.
* Patients with systemic diseases that may affect normal healing.
* Patients with psychiatric problem
* Patients with history of recent radiation therapy to the head and neck area.
* Patients with aggressive periodontitis.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Implant stability evaluation | Immediately after surgery
  Evaluation of implant stability after closed sinus lifting in posterior edentulous maxilla using osteotome technique versus hydraulic lift technique

SECONDARY OUTCOMES:
Patient satisfaction evaluation | Immediately after surgery
  Evaluation of patient satisfaction by using specific numerical questionnaire which depends on numerical scale after closed sinus lifting procedure with implant placement using hydraulic lift technique versus summers' osteotome technique in posterior edentulous maxilla .
  The patient satisfaction numerical questionnaire include several questions to the patient and the patient will put a circle sign on the mark at which he or she feels to represent the answer .
  The numerical scale is from 1 to 5 for each question (with total of 20 questions) :
  1. represents strongly disagree
  2. represents disagree
  3. represents neither agree or disagree
  4. represents agree
  5. represents strongly agree
  The final score is out of 100 so, more higher scores represents more patient satisfaction and so, better outcome and less scores represents less patient satisfaction and so, worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abdelghany, PHD, Principal Investigator — Assoc.professor
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Up till now the strategy of sharing isnot decided